CLINICAL TRIAL: NCT04191200
Title: Etat BUCCO-dentaire de Patients Atteints de SCHIZophrénie et de Troubles Schizo-affectif Suivis au Centre Hospitalier de Charles Perrens
Brief Title: Oral Status of Patients Suffering From SCHIZophrenia Followed at Charles Perrens Hospital
Acronym: BUCCOSCHIZ
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Other Study IDs: BUCCOSCHIZ2019
Record Dates: First submitted 2019-11-28; First posted 2019-12-09 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2019-12

CONDITIONS: Dental Diseases; Schizophrenia
Keywords: Schizophrenia; Psychiatric institutions; Epidemiology; Schizophrenic disorder; Oral Health
MeSH Terms: conditions — Stomatognathic Diseases; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to describe the oral health status of patients suffering from schizophrenia and schizoaffective disorders in a psychiatric institute in France.

DETAILED DESCRIPTION:
Schizophrenia concerns 21 million people in the world and 600 000 in France according to the World Health Organization. This pathology decreases the patient's quality of life and one patient out of two will try to commit suicide and 10% will die. Oral health is an important factor for general well being. The litterature shows that schizophrenic patients tend to visit less dental surgeries than the general population. Patients will often visit the surgery in emergency and dentist often choses to extract instead of a restorative solution. Thus, schizophrenic subjects are 3,4 more likely to become edentulous compared to the general population.

This is a cross-sectional epidemiological study on patients suffering from schizophrenia and and schizoaffective disorders in a psychiatric institution. A dental assessment will be conducted to provide clinical data on oral health. (DMFT, hygiene, mouth dryness, prosthesis) and a survey of their diet, medication, oral quality of life, social security coverage and patients view regarding dental care (Anxiety and Healthcare renunciation).

This is an observational study (oral examination and survey), so no treatment will be compared. The oral health status will be evaluated during one single oral examination and survey during the patient's stay at hospital.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenic patients and patients with schizoaffective disorders at the Charles Perrens Hospital
* Willing to participate in the study
* 18 years old and above

Exclusion Criteria:

* Patients mentally unable to participate or refusing to participate in this study.
* Patient hospitalized under duress
* Minor
* Patients unable to read, speak or write French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Schizophrenic adults and adults with schizoaffective disorders at the Charles Perrens Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Measure of the number of caries, fillings and teeth missing | 1 day
  The main outcome will be to measure the number of caries, fillings and teeth missing as stated in the DMFT Index.
Evaluation of oral hygiene | 1 day
  Oral hygiene will be measured with the simplified oral hygiene index (OHI-S)
Assessement of temporo mandibular dysfunction | 1 day
  Number of patients suffering from temporo mandibular dysfunction (for patients who have replied yes to the 3Q/TMD screening).
Assessing of mouth dryness | 1 day
  Assessing mouth dryness through the Xerostomia Inventory survey.

SECONDARY OUTCOMES:
Link between quality of life and oral health: survey | 1 day
  - Assessment of the link between quality of life and oral health through the GOHAI survey.
Social security coverage | 1 day
  Number of patients and kind of social security coverage
Reason for primary appointment | 1 day
  Assessment for primary reason appointment and dental anxiety measured through the modified dental anxiety scale (MDAS).
Measurement of dental anxiety | 1 day
  Measurement of dental anxiety through the modified dental anxiety scale (MDAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier CHARLES PERRENS, Bordeaux, France

REFERENCES:
- [Background] Denis F. [The oral health of patients in psychiatric institutions and related comorbidities]. Soins Psychiatr. 2014 Jan-Feb;(290):40-4. French. PMID 24620549
- [Background] Curien R. & al; Evaluation de l'influence des psychotropes sur la santé bucco-dentaire chez une population de patients hospitalisés en secteur psychiatrique. Information Dentaire. 88 : (2006): 439-441
- [Background] Bertaud-Gounot V, Kovess-Masfety V, Perrus C, Trohel G, Richard F. Oral health status and treatment needs among psychiatric inpatients in Rennes, France: a cross-sectional study. BMC Psychiatry. 2013 Sep 21;13:227. doi: 10.1186/1471-244X-13-227. PMID 24053587
- [Background] Catteau C, Blaizot A, Duhamel A, Delzenne A, Devillers A, Frimat P. [Dental status and related factors in an occupational health service in Northern France]. Sante Publique. 2013 Nov-Dec;25(6):747-55. French. PMID 24451420